CLINICAL TRIAL: NCT01364090
Title: A Phase IV, Open-label, Multicentre, International Trial of Response Guided Treatment With Directly Observed Pegylated Interferon Alfa 2b (PEG-IFN-alfa 2b) and Self Administered Ribavirin (RBV) for Patients With Chronic HCV Genotype 2 or 3 and Injection Drug Use
Brief Title: A Collaborative Trial in Injectors of Individualized Treatment for Genotype 2/3
Acronym: ACTIVATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1007
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C; treatment; injection drug users or receiving opiate substitution therapy
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment Duration (24 weeks) (Active Comparator): Subjects with detectable HCV RNA after four weeks of therapy will continue on PEG-IFN and ribavirin until week 24 and follow-up for an additional 24 weeks following treatment completion (48 weeks in total).
  Interventions: Drug: Pegylated interferon alfa 2b; Drug: Ribavirin
- Shortened Treatment Duration (12 Weeks) (Experimental): Subjects with undetectable HCV RNA after four weeks of therapy will continue on PEG-IFN and ribavirin until week 12 and follow-up for an additional 24 weeks following treatment completion (36 weeks in total).
  Interventions: Drug: Pegylated interferon alfa 2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa 2b — Pegylated interferon alfa 2b 1.5 mcg/kg/week to a maximum of 150 mcg/week administered subcutaneously once weekly directly observed.
  Other Names: PegInteron
Drug: Ribavirin — Ribavirin - 800-1400 mg daily according to weight taken orally with food, self administered in split doses.

SUMMARY:
This sudy will determine whether shortening treatment for hepatitis C is feasible, safe and effective for patients who are current injection drug users or receiving opiate substitution therapy and who are responding well to treatment early on.

DETAILED DESCRIPTION:
The study will evaluate the feasibility, safety and effectiveness of shortened treatment for hepatitis C genotypes 2/3 in current injection drug users or receiving opiate substitution therapy. Treatment will be with pegylated interferon alfa 2b (directly observed) and ribavirin for 12 weeks in those that have non-quantifiable (<15 IU/ml detected and <15 IU/ml undetected) HCV RNA or undetectable HCV RNA on qualitative assay at week 4 and 24 weeks in those that have quantifiable (≥15 IU/ml) HCV RNA or detectable HCV RNA on qualitative assay at week 4.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* chronic HCV infection
* HCV genotype 2/3 infection
* active injection drug use (within 24 weeks prior to consent) or currently receiving opiate substitution therapy
* compensated liver disease
* negative pregnancy test (within 24 hours of first dose of study medication)
* effective contraception for the duration of the study
* written informed consent

Exclusion Criteria:

* previous interferon or ribavirin therapy
* investigation drug use in the 6 weeks prior to first dose of study medication
* infection with HCV genotypes other than 2/3
* HIV infection
* HBV infection
* ongoing severe psychiatric disease
* frequent drug use that is judged by the treating physician to compromise treatment safety
* standard clinical and medical exclusions for treatment with pegylated interferon alfa 2b and ribavirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Dore, MBBS, PhD, Study Chair — University of New South Wales; Olav Dalgard, MD PhD, Study Chair — University Hospital, Akershus
Locations (17):
- Australia (5):
  - Hunter Pharmacotherapy, Newcastle, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Alfred Hospital, Melbourne, Victoria
- Belgium (2):
  - ZNA Stuivenberg / MSOC Free Clinic, Antwerp
  - Ziekenhuis Oost Limburg / MSOC Limburg, Genk
- Canada (3):
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - East Toronto Hepatitis C Program, Toronto, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- Praxiszentrum Im Tal (PIT), Munich, Germany
- Oslo/Akershus University hospitals, Oslo, Lorenskog, Norway
- Switzerland (3):
  - Basel Zentrum fur Suchtmedizin, Basel
  - Koda Bern/Poliklinik fur Infektiologe, Bern
  - ARUD, Poliklinik Zokl 1, Zurich
- United Kingdom (2):
  - East London Foundation NHS Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] Cunningham EB, Hajarizadeh B, Dalgard O, Amin J, Hellard M, Foster GR, Bruggmann P, Conway B, Backmund M, Robaeys G, Swan T, Marks PS, Quiene S, Applegate TL, Weltman M, Shaw D, Dunlop A, Bruneau J, Midgard H, Bourgeois S, Thurnheer MC, Dore GJ, Grebely J; ACTIVATE Study Group. Adherence to response-guided pegylated interferon and ribavirin for people who inject drugs with hepatitis C virus genotype 2/3 infection: the ACTIVATE study. BMC Infect Dis. 2017 Jun 13;17(1):420. doi: 10.1186/s12879-017-2517-3. PMID 28610605

RESULTS

PARTICIPANT FLOW:
Groups:
- Shortened Treatment Duration (12 Weeks): Subjects with undetectable HCV RNA after four weeks of therapy will continue on pegylated interferon alfa 2b (PEG-IFN) and ribavirin (RBV) until week 12 and follow-up for an additional 24 weeks following treatment completion (36 weeks in total).
  Pegylated interferon alfa 2b: Pegylated interferon alfa 2b 1.5 mcg/kg/week to a maximum of 150 mcg/week administered subcutaneously once weekly directly observed.
  Ribavirin: Ribavirin - 800-1400 mg daily according to weight taken orally with food, self administered in split doses.
- Standard Treatment Duration (24 Weeks): Subjects with detectable HCV RNA after four weeks of therapy will continue on pegylated interferon alfa 2b (PEG-IFN) and ribavirin (RBV) until week 24 and follow-up for an additional 24 weeks following treatment completion (48 weeks in total).
  Pegylated interferon alfa 2b: Pegylated interferon alfa 2b 1.5 mcg/kg/week to a maximum of 150 mcg/week administered subcutaneously once weekly directly observed.
  Ribavirin: Ribavirin - 800-1400 mg daily according to weight taken orally with food, self administered in split doses.
- Discontinued Prior to Week 4: Participants who discontinued therapy prior to week 4 HCV RNA assessment and were therefore not placed in either study arms.
Period: Overall Study
Arm/Group | Shortened Treatment Duration (12 Weeks) | Standard Treatment Duration (24 Weeks) | Discontinued Prior to Week 4
Started | 61 | 26 | 6
Completed | 58 | 12 | 0
Not Completed | 3 | 14 | 6

BASELINE CHARACTERISTICS:
Groups:
- Discontinued Prior to RVR: Participants who discontinued therapy prior to RVR assessment at week 4 and were therefore not placed in either study arms.
- Total: Total of all reporting groups
Arm/Group | Standard Treatment Duration (24 Weeks) | Shortened Treatment Duration (12 Weeks) | Discontinued Prior to RVR | Total
Number analyzed (Participants) | 26 | 61 | 6 | 93
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [35 to 48] | 41 [34 to 49] | 50 [41 to 56] | 41 [35 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 1 | 16
  Male | 23 | 49 | 5 | 77

OUTCOME MEASURES:

1. Primary Outcome: Treatment Efficacy
Description: The primary outcome measure is the number of patients with undetectable HCV RNA at 12 weeks post end of treatment (SVR12) following directly observed PEG-IFN alfa-2b in combination with self-administered ribavirin for 12 weeks in participants with non-quantifiable (<15 IU/ml detected and <15 IU/ml undetected) HCV RNA or undetectable HCV RNA on qualitative assay at week 4 of therapy and for 24 weeks in participants with quantifiable (≥15 IU/ml) HCV RNA or detectable HCV RNA on qualitative assay at week 4 of therapy.
Time Frame: 36 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Duration (24 Weeks) | Shortened Treatment Duration (12 Weeks) | Discontinued Prior to RVR
Number analyzed (Participants) | 26 | 61 | 6
Participants | 10 | 51 | 0

2. Secondary Outcome: Treatment Adherence
Description: Evaluate the adherence (>80 of PEG-IFN, >80% of RBV, >80% of time) to directly observed PEG-IFN alfa-2b in combination with self-administered ribavirin for 12 weeks in participants with non-quantifiable HCV RNA or undetectable HCV RNA on qualitative assay at week 4 of therapy and for 24 weeks in participants with quantifiable HCV RNA or detectable HCV RNA on qualitative assay at week 4 of therapy.
Time Frame: 48 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Treatment Response (ETR & SVR24)
Description: Evaluate the percentage with undetectable HCV RNA at end of treatment (ETR) and 24 weeks post end of treatment (SVR24) in participants treated with PEG-IFN alfa-2b in combination with self-administered ribavirin for 12 weeks in participants with non quantifiable HCV RNA or undetectable HCV RNA at week 4 of therapy and for 24 weeks in participants with quantifiable HCV RNA or detectable HCV RNA at week 4 of therapy.
Time Frame: 48 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Behavioral and Quality of Life
Description: Evaluate changes in illicit drug use, opiate substitution therapy, depression, suicidal ideations and health-related quality of life in participants treated with PEG-IFN alfa-2b in combination with self-administered ribavirin for 12 weeks in participants with non-quantifiable HCV RNA or undetectable HCV RNA on qualitative assay at week 4 of therapy and for 24 weeks in participants with quantifiable HCV RNA or detectable HCV RNA at week 4 of therapy.
Time Frame: 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of signing the consent until 24 weeks post-treatment.
Description: Laboratory abnormalities only recorded as AEs if it caused a Serious Adverse Event (SAE), resulted in discontinuation/modification of study treatment or required treatment with, or modification to, concomitant medication. Pre-existing conditions/diseases that occurred during the study were not considered as adverse events unless they changed in frequency or severity. Participants were assessed at each study visit for adverse events.
Arm/Group | Standard Treatment Duration (24 Weeks) | Shortened Treatment Duration (12 Weeks) | Discontinued Prior to RVR
Serious Adverse Events (participants affected / at risk) | 4/26 | 6/61 | 1/6
Other Adverse Events (participants affected / at risk) | 26/26 | 60/61 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment Duration (24 Weeks) (N=26) | Shortened Treatment Duration (12 Weeks) (N=61) | Discontinued Prior to RVR (N=6)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Treatment Duration (24 Weeks) (N=26) | Shortened Treatment Duration (12 Weeks) (N=61) | Discontinued Prior to RVR (N=6)
Fatigue (General disorders) | 14 | 33 | 1
Influenza like illness (General disorders) | 13 | 19 | 4
Headache (Nervous system disorders) | 14 | 21 | 0
Nausea (Gastrointestinal disorders) | 5 | 26 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 18 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 19 | 0
Insomnia (Psychiatric disorders) | 4 | 15 | 0
Vomiting (Gastrointestinal disorders) | 5 | 11 | 2
Anaemia (Blood and lymphatic system disorders) | 5 | 12 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 5 | 12 | 0
Injection site erythema (General disorders) | 4 | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No